CLINICAL TRIAL: NCT00017225
Title: Neuroblastoma Study Phase II Study of Various Therapies in Patients With Neuroblastoma
Brief Title: Chemotherapy and Radiation Therapy With or Without Peripheral Stem Cell Transplantation in Treating Patients With Neuroblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: German Society for Pediatric Oncology and Hematology GPOH gGmbH (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: GPOH-GERMANY-NB97; CDR0000068664 (Registry Identifier: PDQ (Physician Data Query)); EU-20102; GER-GPOH-NB97
Record Dates: First submitted 2001-06-06; First posted 2003-01-27 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2002-08

CONDITIONS: Neuroblastoma
Keywords: localized resectable neuroblastoma; regional neuroblastoma; disseminated neuroblastoma; stage 4S neuroblastoma; recurrent neuroblastoma; localized unresectable neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — Filgrastim; Carboplatin; Cisplatin; Cyclophosphamide; Dacarbazine; Doxorubicin; Etoposide; Ifosfamide; Melphalan; Tretinoin; Vincristine; Vindesine; Peripheral Blood Stem Cell Transplantation; Radiotherapy

INTERVENTIONS:
Biological: filgrastim
Drug: carboplatin
Drug: cisplatin
Drug: cyclophosphamide
Drug: dacarbazine
Drug: doxorubicin hydrochloride
Drug: etoposide
Drug: ifosfamide
Drug: melphalan
Drug: tretinoin
Drug: vincristine sulfate
Drug: vindesine
Procedure: autologous bone marrow transplantation
Procedure: conventional surgery
Procedure: peripheral blood stem cell transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Peripheral stem cell transplantation may be able to replace immune cells that were destroyed by chemotherapy or radiation therapy used to kill tumor cells. Combining these therapies may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining chemotherapy and radiation therapy with or without peripheral stem cell transplantation in treating patients who have neuroblastoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the frequency of spontaneous remission in pediatric patients with localized neuroblastoma.
* Determine the course of regression in patients with spontaneous remission.
* Determine the event-free survival rate of patients with high-risk neuroblastoma treated with maintenance chemotherapy OR consolidation chemotherapy followed by autologous stem cell rescue.
* Determine if a correlation exists between long-term overall survival and catecholamine response in these high-risk patients.
* Determine if a correlation exists between cytotoxic and conditioning chemotherapies, in terms of bone marrow toxicity, in these high-risk patients.

OUTLINE: This is a multicenter study. Patients are stratified according to risk (low vs standard vs high).

* Observation stratum (low risk): Patients undergo surgical biopsy followed by observation for 6-12 months. Patients may also undergo second-look surgery. Patients with tumor regression receive no further therapy. Patients with disease progression or no tumor regression receive standard-risk chemotherapy as in the standard-risk stratum.
* Standard-risk stratum: Patients undergo surgical biopsy. Patients at least 6 months of age receive 1 course of chemotherapy comprising cisplatin IV and etoposide IV continuously on days 1-4 and vindesine IV over 1 hour on day 1. Patients then receive 1 course of chemotherapy comprising vincristine IV over 1 hour on days 1 and 8, dacarbazine IV over 1 hour on days 1-5, ifosfamide IV continuously on days 1-5, and doxorubicin IV over 4 hours on days 6 and 7.

Patients under 6 months of age receive doxorubicin IV over 30 minutes and vincristine IV on days 1, 3, and 5 and cyclophosphamide IV over 5 minutes on days 1-7. Treatment repeats every 3 weeks for 2 courses in the absence of unacceptable toxicity.

After chemotherapy, patients may undergo second-look surgery followed by 2 additional courses of chemotherapy as above. Patients with complete response or very good partial response receive no further therapy. Patients with partial response, minimal response, no response, or progressive disease undergo local radiotherapy daily 5 days a week for approximately 6 weeks. Patients with no response after radiotherapy may then receive therapy as in the high-risk stratum.

* High-risk stratum: Patients undergo surgical biopsy. Patients at least 6 months of age receive induction chemotherapy comprising cisplatin, etoposide, and vindesine as in the standard-risk stratum combined with filgrastim (G-CSF) subcutaneously (SC) daily beginning on day 8 and continuing until blood counts recover. Patients also receive alternating courses of vincristine, dacarbazine, ifosfamide, and doxorubicin as in the standard-risk stratum combined with G-CSF SC daily beginning on day 9 and continuing until blood counts recover. Treatment repeats every 3 weeks for up to 6 courses in the absence of unacceptable toxicity.

Patients under 6 months of age receive 2 courses of induction chemotherapy as in the standard-risk stratum followed by 4 courses of alternating chemotherapy as above.

Patients may also undergo second-look surgery.

Patients then receive consolidation chemotherapy comprising melphalan IV over 30 minutes on days -8 to -5, etoposide IV over 4 hours on day -4, and carboplatin IV over 1 hour on days -4 to -2. Patients undergo autologous stem cell transplantation (ASCT) on day 0. Patients also receive G-CSF SC or IV over 2 hours daily beginning on day 0. Patients may then undergo radiotherapy daily 5 days a week for 6 weeks.

Patients who were diagnosed less than 1 year ago and who do not demonstrate MYCN amplication receive maintenance chemotherapy comprising oral cyclophosphamide on days 1-8 (instead of consolidation chemotherapy and ASCT as above). Treatment repeats every 3 weeks for 4 courses.

Beginning 4-6 weeks after transplantation or 4 weeks after initiation of the last course of maintenance chemotherapy, all patients receive consolidation therapy with oral tretinoin 3 times daily on days 1-14. Treatment repeats every 28 days for 6 courses followed by a 3-month rest. Patients then receive 3 additional courses.

Patients are followed at 6 weeks, every 3 months for 5 years, and then every 6 months thereafter.

PROJECTED ACCRUAL: Approximately 130 patients (50 in high-risk stratum, 15 in standard-risk stratum, and 65 in observation stratum) will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed neuroblastoma
* Observation stratum:

  * MYCN gene not amplified
  * Infants with stage I-IVS disease OR
  * Over 1 year of age and stage I or II resectable disease
* Standard-risk stratum:

  * MYCN gene not amplified
  * Infants with serious symptoms and stage II-IVS disease OR
  * Over 1 year of age with stage II or III unresectable disease
* High-risk stratum:

  * Stage IV disease OR
  * Stage I-IVS MYCN gene-amplified disease

PATIENT CHARACTERISTICS:

Age:

* 20 and under

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* No kidney insufficiency

Cardiovascular:

* No cardiac insufficiency

Other:

* Not pregnant
* Fertile patients must use effective contraception
* No other serious illness

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy within 6 months after diagnosis

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 1997-05; Study Completion 2002-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Berthold, MD, Study Chair — Children's Hospital Medical Center, Cincinnati
Locations (94):
- Germany (89):
  - Urologische Klinik - Universitaetsklinikum Aachen, Aachen
  - Kinderkrankenhaus Josefinum, Augsburg
  - Zentralklinikum Augsburg, Augsburg
  - Caritaskrankenhaus, Bad Mergentheim
  - Klinikum Bayreuth, Bayreuth
  - Helios Klinikum Berlin, Berlin
  - Charite - Campus Virchow Klinikum, Berlin
  - Krankenanstalten Gilead, Biefeld
  - Kinderklinik der Universitaet-Bonn, Bonn
  - Stadt Klinikum - Howedestrase, Braunschweig
  - Zentralkrankenhaus, Bremen
  - Klinikum Chemnitz GMBH, Chemnitz
  - Klinikum Coburg, Coburg
  - Medizinische Universitaetsklinik I, Cologne
  - Carl - Thiem - Klinkum Cottbus, Cottbus
  - Vestische Kinderklinik, Datteln
  - Klinikum Lippe - Detmold, Detmold
  - Stadt. Kliniken, Dortmund
  - Stadt. KH Dresden - Neustadt, Dresden
  - Universitatsklinikum Carl Gustav Carl Carus, Dresden
  - Universitaetsklinik Duesseldorf, Düsseldorf
  - Helios Klinikum Erfurt GmbH, Erfurt
  - Universitaets - Kinderklinik, Erlangen
  - Universitaetsklinikum Essen, Essen
  - Klinikum der J.W. Goethe Universitaet, Frankfurt
  - Universitaetskinderklinik - Universitaetsklinikum Freiburg, Freiburg im Breisgau
  - Stadt. Kinderklinik, Gelsenkirchen
  - Kinderklinik, Giessen
  - Universitaetsklinikum Goettingen, Göttingen
  - Universitats - Kinderklinik, Greiswald
  - Kreiskrankenhaus Gummersbach GMBH, Gummersbach
  - St. Barbara Krankenhaus, Halle
  - Martin Luther Universitaet, Halle
  - Altonaer Kinderkrankenhaus, Hamburg
  - Universitaets-Krankenhaus Eppendorf, Hamburg
  - Evangelische Krankenhaus Hamm, Hamm
  - Kinderkrankenhaus auf der Bult, Hanover
  - Medizinische Hochschule Hannover, Hanover
  - Universitaets-Kinderklinik Heidelberg, Heidelberg
  - Gemeinschaftskrankenhaus, Herdecke
  - Universitatsklinik Homburg, Homburg
  - Marien Hospital, Homburg
  - Praxis am Evangelischen Krankenhaus Bethanien, Iserlohn
  - Universitaets - Kinderklinik, Jena
  - Westpfalz-Klinikum GmbH, Kaiserslautern
  - Stadt. Kinderklinik, Karlsruhe
  - Kinderkrankenhaus, Kassel
  - Klinikum Kassel, Kassel
  - Staedtische Krankenhaus Kiel, Kiel
  - University Hospital Schleswig-Holstein - Kiel Campus, Kiel
  - Stadt. Krankenhaus Kemperhof, Koblenz
  - Staedtisches Kinderkrankenhaus, Koln - Riehl
  - Klinik Konstanz, Konstanz
  - Klinikum Krefeld GmbH, Krefeld
  - Universitaets - Kinderklinik, Leipzig
  - Universitaets Klinik fuer Kinderchirurgie, Leipzig
  - St. Annastift Krankenhaus, Ludwigshafen
  - Universitaets - Kinderklinik - Luebeck, Lübeck
  - Universitatsklinikum der MA, Magdeburg
  - Johannes Gutenberg University, Mainz
  - Stadt. Klinik - Kinderklinik, Mannheim
  - Universitaets - Kinderklinik, Marburg
  - Klinikum Minden, Minden
  - Universitaets - Kinderpoliklinik, Munich
  - Kinderklinik d. TU / Schwabing, Munich
  - Staedtisches Krankenhaus Muenchen - Harlaching, Munich
  - Kinderklinik, Munich
  - Klinik und Poliklinik fuer Kinderheilkunde - Universitaetsklinikum Muenster, Münster
  - Kinderklinik Kohlhof, Neunkirchen
  - Cnopfche Kinderklinik, Nuremberg
  - Klinikum Oldenburg, Oldenburg
  - Kindershospital, Osnabrück
  - Krankenhaus D Barmherzigen Brueder, Regensburg
  - Staedtische Klinikum-Kinderklinik, Rosenheim
  - Kinderklinik - Universitaetsklinikum Rostock, Rostock
  - Saarbrucker Winterbergkliniken, Saarbrücken
  - Johanniter-Kinderklinik, Sankt Augustin
  - Diakone - Krankenhaus, Schwäbisch Hall
  - Klinikum Schwerin, Schwerin
  - Leopoldina - Krankenhaus, Schwienfurt
  - Deutsches Rotes Kreuz, Siegen
  - Olgahospital, Stuttgart
  - Mutterhaus der Borromaerinnen, Trier
  - Universitaetsklinikum Tuebingen, Tübingen
  - Universitaet Ulm, Ulm
  - St. Marien Hospital, Vechta
  - Reinhard - Nieter - Krankenhaus, Wilhelmshaven
  - Helios Klinikum Wuppertal, Wuppertal
  - Universitaets - Kinderklinik Wuerzburg, Würzburg
- Academisch Ziekenhuis Maastricht, Maastricht, Netherlands
- Switzerland (4):
  - University Children's Hospital, Basel
  - Ospedale "la Carita", Locarno, Locarno
  - Kinderspital Luzerne, Luzerne 16
  - University Children's Hospital, Zurich

REFERENCES:
- [Background] Krams M, Hero B, Berthold F, Parwaresch R, Harms D, Rudolph P. Proliferation marker KI-S5 discriminates between favorable and adverse prognosis in advanced stages of neuroblastoma with and without MYCN amplification. Cancer. 2002 Feb 1;94(3):854-61. PMID 11857322
- [Background] Simon T, Hero B, Dupuis W, Selle B, Berthold F. The incidence of hearing impairment after successful treatment of neuroblastoma. Klin Padiatr. 2002 Jul-Aug;214(4):149-52. doi: 10.1055/s-2002-33179. PMID 12165893
- [Background] Spitz R, Hero B, Westermann F, Ernestus K, Schwab M, Berthold F. Fluorescence in situ hybridization analyses of chromosome band 1p36 in neuroblastoma detect two classes of alterations. Genes Chromosomes Cancer. 2002 Jul;34(3):299-305. doi: 10.1002/gcc.10070. PMID 12007190
- [Background] Hero B, Simon T, Spitz R, Ernestus K, Gnekow AK, Scheel-Walter HG, Schwabe D, Schilling FH, Benz-Bohm G, Berthold F. Localized infant neuroblastomas often show spontaneous regression: results of the prospective trials NB95-S and NB97. J Clin Oncol. 2008 Mar 20;26(9):1504-10. doi: 10.1200/JCO.2007.12.3349. PMID 18349403
- [Background] Simon T, Hero B, Benz-Bohm G, von Schweinitz D, Berthold F. Review of image defined risk factors in localized neuroblastoma patients: Results of the GPOH NB97 trial. Pediatr Blood Cancer. 2008 May;50(5):965-9. doi: 10.1002/pbc.21343. PMID 17914735
- [Background] Berthold F, Hero B, Kremens B, Handgretinger R, Henze G, Schilling FH, Schrappe M, Simon T, Spix C. Long-term results and risk profiles of patients in five consecutive trials (1979-1997) with stage 4 neuroblastoma over 1 year of age. Cancer Lett. 2003 Jul 18;197(1-2):11-7. doi: 10.1016/s0304-3835(03)00076-4. PMID 12880954
- [Background] Spitz R, Hero B, Ernestus K, Berthold F. Deletions in chromosome arms 3p and 11q are new prognostic markers in localized and 4s neuroblastoma. Clin Cancer Res. 2003 Jan;9(1):52-8. PMID 12538451
- [Background] Spitz R, Hero B, Ernestus K, Berthold F. FISH analyses for alterations in chromosomes 1, 2, 3, and 11 define high-risk groups in neuroblastoma. Med Pediatr Oncol. 2003 Jul;41(1):30-5. doi: 10.1002/mpo.10313. PMID 12764740
- [Background] Spitz R, Hero B, Ernestus K, Berthold F. Gain of distal chromosome arm 17q is not associated with poor prognosis in neuroblastoma. Clin Cancer Res. 2003 Oct 15;9(13):4835-40. PMID 14581355
- [Background] von Schweinitz D, Hero B, Berthold F. The impact of surgical radicality on outcome in childhood neuroblastoma. Eur J Pediatr Surg. 2002 Dec;12(6):402-9. doi: 10.1055/s-2002-36952. PMID 12548494
- [Result] Simon T, Hero B, Bongartz R, Schmidt M, Muller RP, Berthold F. Intensified external-beam radiation therapy improves the outcome of stage 4 neuroblastoma in children > 1 year with residual local disease. Strahlenther Onkol. 2006 Jul;182(7):389-94. doi: 10.1007/s00066-006-1498-8. PMID 16826357
- [Result] Kremens B, Hero B, Esser J, Weinel P, Filger-Brillinger J, Fleischhack G, Graf N, Gruttner HP, Niemeyer C, Schulz A, Wickmann L, Berthold F. Ocular symptoms in children treated with human-mouse chimeric anti-GD2 mAb ch14.18 for neuroblastoma. Cancer Immunol Immunother. 2002 Apr;51(2):107-10. doi: 10.1007/s00262-001-0259-x. Epub 2002 Feb 1. PMID 11904735
- [Derived] Decarolis B, Simon T, Krug B, Leuschner I, Vokuhl C, Kaatsch P, von Schweinitz D, Klingebiel T, Mueller I, Schweigerer L, Berthold F, Hero B. Treatment and outcome of Ganglioneuroma and Ganglioneuroblastoma intermixed. BMC Cancer. 2016 Jul 27;16:542. doi: 10.1186/s12885-016-2513-9. PMID 27465021